CLINICAL TRIAL: NCT00012220
Title: A Randomized Phase II Study Of Gemcitabine/Cisplatin, Gemcitabine/Docetaxel, Gemcitabine/Irinotecan, Or Fixed Dose Rate Infusion Gemcitabine In Patients With Metastic Pancreatic Cancer
Brief Title: Gemcitabine Alone or in Combination With Other Chemotherapy Drugs in Treating Patients With Metastatic Cancer of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-89904; U10CA031946 (NIH); CALGB-89904; CDR0000068495 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cisplatin; Docetaxel; Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Gemcitabine (Active Comparator): Standard treatment
  Interventions: Drug: gemcitabine hydrochloride
- Gemcitabine + cisplastin (Experimental): Addition of cisplastin to gemcitabine
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride
- Gemcitabine + docetaxel (Experimental): Addition of docetaxel to gemcitabine
  Interventions: Drug: docetaxel; Drug: gemcitabine hydrochloride
- Gemcitabine + Irinotecan (Experimental): Addition of irinotecan to gemcitabine
  Interventions: Drug: gemcitabine hydrochloride; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: cisplatin — 50 mg/sq m IV infusion over 30 min on Days 1 & 15 of ea cycle
  Arms: Gemcitabine + cisplastin
Drug: docetaxel — 40 mg/sq m IV infusion over 60 min on Days 1 & 8 of ea treatment cycle
  Arms: Gemcitabine + docetaxel
Drug: gemcitabine hydrochloride — Gemcitabine only arm: 1500 mg/sq m in 250 mL NS IV infusion over 150 min Days 1, 8, & 15 of ea cycle
  * cisplastin arm: 1000 mg/sq m 250 mL NS IV infusion over 30 min Days 1, 8, 15 of ea cycle
  * docetaxel and + irinotecan arms: 1000 mg/sq m in 250 mL NS IV infusion over 30 min Days 1 & 8 of ea cycle
Drug: irinotecan hydrochloride — 100 mg/q m in 500 mL D5W or D5NS IV infusion over 90 min Days 1 & 8 of ea cycle
  Arms: Gemcitabine + Irinotecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if gemcitabine is more effective when given alone or in combination with another chemotherapy drug in treating cancer of the pancreas.

PURPOSE: Randomized phase II trial to compare the effectiveness of gemcitabine given alone or in combination with other chemotherapy drugs in treating patients who have metastatic cancer of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival rate of patients with metastatic pancreatic cancer treated with gemcitabine alone vs with cisplatin vs with docetaxel vs with irinotecan.
* Compare the time to disease progression in patients treated with these regimens.
* Compare the CA 19-9 biomarker response in patients treated with these regimens.
* Correlate the CA 19-9 biomarker response with survival in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the response in patients with measurable disease treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of four treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 followed by cisplatin IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine IV over 150 minutes on days 1, 8, and 15. Treatment repeats every 28 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.
* Arm III: Patients receive gemcitabine IV over 30 minutes followed by docetaxel IV over 60 minutes on days 1 and 8. Treatment repeats every 21 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.
* Arm IV: Patients receive gemcitabine IV over 30 minutes followed by irinotecan IV over 90 minutes on days 1 and 8. Treatment repeats every 21 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 240 patients (60 per arm) will be accrued for this study within 30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas
* Metastatic disease by CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* CTC 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 2.5 times ULN if SGOT greater than 1.5 times ULN
* Alkaline phosphatase any value if SGOT less than 1.5 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study
* No other currently active malignancy (completed therapy and considered to be at less than 30% risk of relapse) except non-melanoma skin cancer

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* No prior chemotherapy except fluorouracil (5-FU)
* At least 2 weeks since prior 5-FU
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except steroids for adrenal failure, hormonal therapy for non-disease related conditions (e.g., insulin for diabetes), or intermittent use of dexamethasone as an antiemetic

Radiotherapy:

* At least 2 weeks since prior radiotherapy
* No concurrent palliative radiotherapy except whole-brain irradiation for CNS disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2001-01; Primary Completion 2004-06 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 4 years post treatment

SECONDARY OUTCOMES:
Time to disease progression | treatment up to 4 years post treatment
Toxicity | treatment and up to 4 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kulke, MD, Study Chair — Dana-Farber Cancer Institute
Locations (76):
- United States (75):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Helen and Harry Gray Cancer Institute at Good Samaritan Medical Center, West Palm Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Result] Kulke MH, Tempero MA, Niedzwiecki D, Hollis DR, Kindler HL, Cusnir M, Enzinger PC, Gorsch SM, Goldberg RM, Mayer RJ. Randomized phase II study of gemcitabine administered at a fixed dose rate or in combination with cisplatin, docetaxel, or irinotecan in patients with metastatic pancreatic cancer: CALGB 89904. J Clin Oncol. 2009 Nov 20;27(33):5506-12. doi: 10.1200/JCO.2009.22.1309. Epub 2009 Oct 26. PMID 19858396